CLINICAL TRIAL: NCT03720158
Title: Effect of Enteral Supplementation of Omega 3 Fatty Acids on the Quality of Life and Functionality of Patients With Head and Neck Squamous Cell Carcinoma Undergoing Radiotherapy
Brief Title: Enteral Omega 3 During Radiotherapy to Improve the Quality of Life and Functionality of Head and Neck Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The activities in the study hospital were seriously impacted by the medical care of COVID patients, affecting the medical management protocol of the study population. This situation does not allow to continue with the recruitment of patients.
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2017-785-110
Record Dates: First submitted 2018-10-15; First posted 2018-10-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Quality of Life; Radiotherapy; Complications
Keywords: Head and Neck Neoplasms; Omega 3 PolyUnsaturated Fatty Acid (PUFA); Quality of Life; Radiotherapy; Cancer Cachexia
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega 3 Group (Experimental): Five mL of an Omega-3 highly concentrated substance (containing 2.25 g of EPA and 1.08 g of DHA) will be added daily to the standard enteral diet during the entire radiotherapy treatment period (from 5-7 weeks)
  Interventions: Dietary Supplement: Omega 3 Group
- Placebo or Control Group (Placebo Comparator): Five mL of pigmented and flavored corn oil will be added daily to the standard enteral diet during the entire radiotherapy treatment period (from 5-7 weeks)
  Interventions: Dietary Supplement: Placebo or Control Group

INTERVENTIONS:
Dietary Supplement: Omega 3 Group — Five mL of an Omega-3 highly concentrated substance (containing 2.25 g of EPA and 1.08 g of DHA) will be added daily to the standard enteral diet during the entire radiotherapy
  Other Names: Enteral administration of Omega 3 Fatty Acids
  Arms: Omega 3 Group
Dietary Supplement: Placebo or Control Group — Five mL of pigmented and flavored corn oil will be added daily to the standard enteral diet during the entire radiotherapy treatment period (from 5-7 weeks)
  Other Names: Enteral administration of Placebo
  Arms: Placebo or Control Group

SUMMARY:
Health-related Quality of Life (QoL) is a multidimensional construct that allows us to know the patient's perception of well-being, and how this perception is related to their illness and treatment. In clinical research, especially clinical trials, the QoL measurement has become an important element to evaluate. In patients with Head and Neck Squamous Cell Carcinoma (HNSCC), low QoL is associated with Malnutrition (MN), and Cancer Cachexia (CC) is a principal component in its multifactorial etiology. The exacerbated hypercatabolic state of CC is caused by the increase of pro-inflammatory cytokines, Reactive Oxygen Species (ROS), and other catabolic mediators. The clinical manifestation of CC is a continuous decrease in muscle mass (with or without loss of fat mass), which is not entirely reversible with nutritional support and which leads to the functional deterioration of patients. Due to CC, the patients with HNSCC who receive total enteral nutritional support have difficulties in maintaining an optimal nutritional status, and this situation is more frequent during RadioTherapy (RT). An immune-modulator nutrient, Omega-3 fatty acids (O3) have shown efficacy in improving the nutritional and inflammatory parameters of patients with HNSCC; however, little is known about their impact on patients' QoL and Functionality (Fx). Therefore, this clinical trial is proposed to provide information about the usefulness of O3 for improving the Fx and QoL of patients with HNSCC receiving total enteral nutrition during RT.

DETAILED DESCRIPTION:
* Objective: To determine the effect of the daily addition of five mL of an O3 highly concentrated substance (EicosaPentaenoic Acid - EPA: 2.25 g and DocosaHexaenoic Acid - DHA: 1.08 g), to the standard enteral nutrition diet during RT (5-7 weeks), on the Quality of Life (QoL) and Functionality (Fx) of patients with HNSCC.
* Methods: Randomized, double-blinded, controlled clinical trial. Patients with HNSCC (ages ranging from 18-80 years) who will receive total enteral nutrition support through percutaneous endoscopic gastrostomy and RT for the first time will be invited to participate in the study. Exclusion criteria are fish allergy, anticoagulant consumption, any supplement consumption 6 months prior to the experiment, any contraindication to the performance of the body composition analysis using bioelectrical impedance (Bioelectrical Impedance Analysis, BIA) (cardiac pacemaker, any metallic prosthesis, inability to stand, severe edema), or the presence of the mal-absorption syndrome, two or more cancer types, organ dysfunction, immune diseases, or any hospitalization during the 20 days prior to extraction of the blood sample. Patients with the consumption of any other nutritional supplement or diagnosed with any other cancer during the treatment period, or with insufficient or incorrectly processed blood-serum samples will be eliminated. After expressing their willingness to participate via the signing of the informed consent document, 86 patients with HNSCC will be allocated into two groups: The O3 Group will have the addition of 5 mL of an O3 highly concentrated substance containing 2.25 g of EPA and 1.08 g of DHA to the standard enteral diet during RT (5-7 weeks), and the Placebo or Control Group will have the addition of 5 mL of a placebo (pigmented and flavored corn oil) in a similar manner. All patients will be seen every 4 weeks at the Nutrition Support Service for nutritional assessment and counseling, and to receive the enteral nutrition containers (standard polymeric diet). On the same day, a Research Assistant (who will be blinded) will provide the supplements or the placebo. The patients' sociodemographic and clinical information, body composition, albumin, hemoglobin, C-reactive protein, tumor cachexia-related cytokines: IL (Interleukin) 1a, IL-1b, IL-6, IL-8, IFNγ (Interferon gamma), TGF-β (transforming growth factor beta), and TNF-α (Tumor necrosis factor alpha); and responses for the European Organisation for Research and Treatment of Cancer Quality of Life C-30 (EORTC-QLQ-C30) with the Head and Neck Cancer module (EORTC-QLQ-H&N35) questionnaires will be collected at the beginning of RT, at the end of RT, and 12 weeks after starting RT. Statistical analysis includes descriptive statistics, inference statistics (Student t-test, Mann-Whitney test, one-way ANOVA with Bonferroni correction, Kruskal-Wallis with Dunn's non-parametric test), and the Cox regression; an intention-to-treat analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Head and Neck Squamous Cell Carcinoma (HNSCC) confirmed by histologic
* Eligible for receiving total enteral nutrition support through percutaneous endoscopic gastrostomy for the first time
* Eligible for receiving RadioTherapy (RT) for the first time

Exclusion Criteria:

* Allergy to fish
* Consumption of anticoagulants
* Consumption of any supplement 6 months prior to the experiment
* Any contraindication to the performance of the Bioelectrical Impedance Analysis (BIA) (cardiac pacemaker, any metallic prosthesis, inability to stand, severe edema)
* Mal-absorption syndrome
* Two or more cancer types
* Organ dysfunction
* Immune diseases
* Any hospitalization during the 20 days prior to extraction of the blood sample

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Global Health Status/Quality of Life (GHS/QoL) subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30) | From baseline (time 0) up to the ending of RT (from 5-7 weeks) (time 1); from baseline up to 12 weeks (time 2)
  The QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item scales and single-item measures. These include five functional scales (physical, role, emotional, social, and cognitive), three symptom scales (fatigue, nausea and vomiting, and pain), a global health status / QoL scale (GHS/QoL), and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and difficulties). Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." The principle for scoring these scales is the same in all cases: 1. Estimate the average of the items that contribute to the scale; this is the raw score. 2. Use a linear transformation to standardize the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms. A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change in Physical Functioning (PF) subscale of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30) | From baseline (time 0) up to the ending of RT (from 5-7 weeks) (time 1); from baseline up to 12 weeks (time 2)
  The QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item scales and single-item measures. These include the Physical Functioning Scale and four more functional scales (role, emotional, social, and cognitive), three symptom scales (fatigue, nausea and vomiting, and pain), a global health status / QoL scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and difficulties). Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." The method for scoring these scales is: 1. Estimate the average of the items that contribute to the scale; this is the raw score. 2. Use a linear transformation to standardize the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms. A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.

SECONDARY OUTCOMES:
Changes in serum cancer cachexia-related cytokines: IL (Interleukin)-1a, IL-1b, IL-6, IL-8, IFNγ (Interferon gamma), TGF-β (transforming growth factor beta), and TNF-α (Tumor necrosis factor alpha) | From baseline (time 0) up to the ending of RT (from 5-7 weeks) (time 1); from baseline up to 12 weeks (time 2)
  Changes of the serum levels quantified by means of the Enzyme-Linked ImmunoSorbent Assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Luz Ma. Adriana Balderas-Peña, PhD, Study Chair — Unidad de Investigación Biomédica 02, UMAE HE CMNO IMSS
Locations (1):
- Unidad de Investigación Biomédica 02, UMAE HE CMNO IMSS, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perloy A, Maasland DHE, van den Brandt PA, Kremer B, Schouten LJ. Intake of meat and fish and risk of head-neck cancer subtypes in the Netherlands Cohort Study. Cancer Causes Control. 2017 Jun;28(6):647-656. doi: 10.1007/s10552-017-0892-0. Epub 2017 Apr 5. PMID 28382514
- [Background] Righini CA, Timi N, Junet P, Bertolo A, Reyt E, Atallah I. Assessment of nutritional status at the time of diagnosis in patients treated for head and neck cancer. Eur Ann Otorhinolaryngol Head Neck Dis. 2013 Feb;130(1):8-14. doi: 10.1016/j.anorl.2012.10.001. Epub 2012 Dec 20. PMID 23266003
- [Background] Ravasco P, Monteiro-Grillo I, Vidal PM, Camilo ME. Nutritional deterioration in cancer: the role of disease and diet. Clin Oncol (R Coll Radiol). 2003 Dec;15(8):443-50. doi: 10.1016/s0936-6555(03)00155-9. PMID 14689999
- [Background] van Bokhorst-de van der Schueren MA, van Leeuwen PA, Sauerwein HP, Kuik DJ, Snow GB, Quak JJ. Assessment of malnutrition parameters in head and neck cancer and their relation to postoperative complications. Head Neck. 1997 Aug;19(5):419-25. doi: 10.1002/(sici)1097-0347(199708)19:53.0.co;2-2. PMID 9243270
- [Background] Sheth CH, Sharp S, Walters ER. Enteral feeding in head and neck cancer patients at a UK cancer centre. J Hum Nutr Diet. 2013 Oct;26(5):421-8. doi: 10.1111/jhn.12029. Epub 2013 Feb 5. PMID 23379517
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Alshadwi A, Nadershah M, Carlson ER, Young LS, Burke PA, Daley BJ. Nutritional considerations for head and neck cancer patients: a review of the literature. J Oral Maxillofac Surg. 2013 Nov;71(11):1853-60. doi: 10.1016/j.joms.2013.04.028. Epub 2013 Jul 9. PMID 23845698
- [Background] Planas M, Puiggros C, Redecillas S. [Contribution of nutritional support to fight cancer cachexia]. Nutr Hosp. 2006 May;21 Suppl 3:27-36. Spanish. PMID 16768028
- [Background] Murphy BA, Ridner S, Wells N, Dietrich M. Quality of life research in head and neck cancer: a review of the current state of the science. Crit Rev Oncol Hematol. 2007 Jun;62(3):251-67. doi: 10.1016/j.critrevonc.2006.07.005. Epub 2007 Apr 3. PMID 17408963
- [Background] Mulasi U, Vock DM, Kuchnia AJ, Jha G, Fujioka N, Rudrapatna V, Patel MR, Teigen L, Earthman CP. Malnutrition Identified by the Academy of Nutrition and Dietetics and American Society for Parenteral and Enteral Nutrition Consensus Criteria and Other Bedside Tools Is Highly Prevalent in a Sample of Individuals Undergoing Treatment for Head and Neck Cancer. JPEN J Parenter Enteral Nutr. 2018 Jan;42(1):139-147. doi: 10.1177/0148607116672264. Epub 2017 Dec 11. PMID 29505143
- See also: World Health Organization. Estimated crude rate of incident cases, both sexes, worldwide (top 20 cancer sites) in 2012 — http://gco.iarc.fr/today/online-analysis-multi-bars?mode=cancer&mode_population=continents&population=900&sex=0&cancer=29&type=0&statistic=0&prevalence=0&color_palette=default